CLINICAL TRIAL: NCT06346795
Title: Clinical Evaluation of Class II Restorations Made With Highly Filled Flowable Composite Resins
Brief Title: Class II Restorations With High-Filled Flowable Composites
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Merve Gurses, Assistant Proffesor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SelcukC
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Dental Caries; Class II Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G-aenial Universal Injectable (Experimental)
  Interventions: Other: High-filling flowable dental composite
- Grandio Flow (Experimental)
  Interventions: Other: High-filling flowable dental composite
- Clearfil Majesty Flow (Experimental)
  Interventions: Other: High-filling flowable dental composite

INTERVENTIONS:
Other: High-filling flowable dental composite — Class II restorations will be performed with G-aenial Universal Injectable, Grandio Flow, and Clearfil Majesty Flow high-filling flowable composites.

SUMMARY:
In the study, Class II restorations will be performed with G-aenial Universal Injectable (GC/ Tokyo, Japan), Grandio Flow (VOCO/ Germany), and Clearfil Majesty Flow (Kuraray/ Japan) composites will evaluated. Restorations will be assessed according to modified USPHS criteria in 1st week, 6th months, and 12th months from the placement date. The Chi-square test will used for statistical analysis of the difference between the groups, and the Cochran Q test will used for the significance of the difference between time-dependent changes within each group (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

A patient presenting with;

1. over 18 years of age
2. a normal periodontal status and good general health
3. proximal caries that are similar in size to premolar and molar teeth
4. vital teeth
5. teeth in contact with the opposing tooth and subjected to normal occlusal forces
6. attend follow-up appointments

Exclusion Criteria:

1. poor oral hygiene status
2. those with severe or chronic periodontitis
3. absence of adjacent and antagonist teeth
4. potential behavioral problems (e.g. bruxism)
5. allergy to any product used in the study
6. exposure of the pulp during cavity preparation
7. systemically unhealthy
8. pregnant and lactating women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Retention | 7th day, 6th month, 12th month.
  No loss of restorative material
Color match | 7th day, 6th month, 12th month.
  The restoration matches the adjacent tooth structure in color and translucency
Marginal discoloration | 7th day, 6th month, 12th month.
  There is no discoloration anywhere on the margin between the restoration and the tooth structure
Marginal adaptation | 7th day, 6th month, 12th month.
  There is no visible evidence of a crevice along the margin into which the explorer will penetrate
Secondary caries | 7th day, 6th month, 12th month.
  No evidence of secondary caries
Surface texture | 7th day, 6th month, 12th month.
  The surface of the restoration does not have any defects
Anatomical form | 7th day, 6th month, 12th month.
  The restoration is continuous with the existing anatomic form
Postoperative sensitivity | 7th day, 6th month, 12th month.
  No postoperative sensitivity, after the restorative procedure and during the study

CONTACTS AND LOCATIONS:
Overall Officials: Merve Gürses, Principal Investigator — Selcuk University, Faculty of Dentistry, Department of Restorative Dentistry
Locations (1):
- Selcuk University, Faculty of Dentistry, Restorative Dentistry Department, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No